CLINICAL TRIAL: NCT00690157
Title: National Polish Registry of Patients Referred for Heart Transplantation. POLKARD HF
Brief Title: Registry of Patients Referred for Heart Transplantation
Acronym: POLKARD HF
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Ministry of Health, Poland (Other Government)
Responsible Party: Jerzy Korewicki, MD, Professor, Institute of Cardiology Warsaw, Poland
Other Study IDs: POLKARD 1304/IK-AG-K-283/03
Record Dates: First submitted 2008-05-29; First posted 2008-06-04 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Advanced Heart Failure; Heart Transplantation
Keywords: heart failure, prognosis, markers,heart transplantation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Main goal of the study is the risk stratification of patients with advanced heart failure referred for orthotopic heart transplantation (OHT) according to HFSS score, other risk factors and biological markers and verification of their prognostic value in Polish population.

DETAILED DESCRIPTION:
PART I 23.10.2008- 31.12.2005 Creation of the Polish national registry of patients referred for cardiac transplantation and after heart transplantation - including urgency of qualification and prognosis.

Main goal of the study is the risk stratification of patients with advanced heart failure referred for orthotopic heart transplantation (OHT) according to HFSS score, other risk factors and biological markers and verification of their prognostic value in Polish population.

All patients with advanced heart failure referred as potential candidates for OHT in all active transplantation centers were included in the registry.

PART II 1.01.2006 -30.11.2007 Since 2006 only patients which were definitely enlisted on the waiting list for heart transplantation were included in the registry

Clinical and laboratory data were recorded in the internet based form. Clinical data included the etiology of the disease, NYHA class, duration of symptoms pharmacological therapy, left ventricular ejection fraction, Ergospirometric maximal oxygen uptake (V02 max) results and right heart catheterization results , ecg data of leading heart rhythm and QRS duration >=0,12 s and other were stored Sodium ,NTproBNP levels and hs CRP plasma levels were recorded during first 48 hours of hospitalization. All patients were followed in a prospective cohort study until the end point : death or OHT , observations were censored at the end of the study. The urgency of OHT and death data was recorded by information from participating centers and national death registry quarries.

Primary end point : Death for all causes or urgent (UNOS 1) heart transplantation Secondary end point: Death without transplantation Death or heart transplantation

Substudy POLKARD HF registry - genetic polymorphism substudy Study start date 01.04.2004 end 30.10.2007

Study population: All consecutive patients included into POLKARD HF registry, who agreed to participate and signed ICF related to the substudy.

Estimated size 350 - 450 patients.

Aims: To describe the potential impact of selected candidate genes polymorphisms on the heart failure prognosis and the survival of patients after orthotropic heart transplantation

ELIGIBILITY:
Inclusion Criteria:

* men and women aged >10 years with advanced heart failure
* referred as potential candidates for orthotropic heart transplantation

Exclusion Criteria:

* refusal to participate in the registry
* not enlisted for heart transplantation (since 2006)

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced heart failure referred for orthotropic heart transplantation (OHT)
Sampling Method: Non-Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2003-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Death for all causes or urgent heart transplantation | prospective progressive 1 to 48 months

SECONDARY OUTCOMES:
Death without heart transplantation | prospective , progressive 1 to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Marian Zembala, MD,PhD, Prof, Principal Investigator — Śląskie Centrum Chorób Serca,Klinika Kardiochirurgii,ul. Szpitalna 2, 41-800 Zabrze; Jerzy Sadowski, MD,PhD, Prof, Principal Investigator — Collegium Medicum Uniwersytetu Jagiellońskiego,Klinika Chirurgii Serca Naczyń i Transplantologii,ul. Prądnicka 80, 31-202 Kraków; Mirosław Garlicki, MD, PhD, Principal Investigator — Klinika Kardiochirurgii Centralnego Szpitala Klinicznego MSWiA, ul. Wołoska 137, 02-507 Warszawa; Jerzy Korewicki, MD,PhD, Prof, Study Director — Klinika Niewydolności Serca i Transplantologii, Instytut Kardiologii, 04-628 Warszawa ul.Alpejska 42; Aldona Browarek, MD, PhD, Principal Investigator — Klinika Niewydolności Serca i Transplantologii, Instytut Kardiologii, 04-628 Warszawa ul.Alpejska 42
Locations (5):
- Poland (5):
  - Klinika Chirurgii Serca, Naczyń i Transplantologii, Szpital im.Jan Pawłą II, Krakow
  - Klinika Kardiochirurgii CSK MSWiA, Warsaw
  - II Klinika Kardiochirurgii Instytutu Kardiologii, Warsaw
  - Klinika Niewydolności Serca i Transplantologii Instytutu Kardiologii, Warsaw
  - Śląskie Centrum Chorób Serca, Zabrze

REFERENCES:
- [Result] Korewicki J., Browarek A., Zielinski T., Sobieszczanska-Małek M., Piotrowska M., Zembala M., Zakliczynski M., Rozentryt P., Baranska-Kosakowska A., Sadowski J., Przybyłowski P., Milaniak I., Garlicki M.: Prognosis of patients with advanced heart failure referred for heart transplantation data of POLKARD HF 2003-2005.[Rokowanie chorych z ciężką niewydolnością serca, wstępnie kwalifikowanych do przeszczepu serca - na podstawie danych ogólnopolskiego rejestru POLKARD 2003-2005.] Kardiochir. Torakochir. Pol., 2006(3): 308 - 322.
- [Derived] Korewicki J. Cardiac transplantation is still the method of choice in the treatment of patients with severe heart failure. Cardiol J. 2009;16(6):493-9. PMID 19950084
- [Derived] Zielinski T, Sobieszczanska-Malek M, Browarek A, Piotrowska M, Zakliczynski M, Przybylowski P, Roguski K, Sadowski J, Zembala M, Korewicki J; POLKARD HF investigators. The influence of the recipient's body weight on the probability to obtain a heart transplant-POLKARD HF registry. Transplant Proc. 2009 Oct;41(8):3166-70. doi: 10.1016/j.transproceed.2009.08.015. PMID 19857703
- [Derived] Zielinski T, Browarek A, Zembala M, Sadowski J, Zakliczynski M, Przybylowski P, Roguski K, Kosakowska AB, Korewicki J; POLKARD HF investigators. Risk stratification of patients with severe heart failure awaiting heart transplantation-prospective national registry POLKARD HF. Transplant Proc. 2009 Oct;41(8):3161-5. doi: 10.1016/j.transproceed.2009.09.049. PMID 19857702
- [Derived] Zielinski T, Kurjata P, Korewicki J; participants of POLKARD-HF. Prognosis in patients with severe heart failure referred for heart transplantation--POLKARD-HF 2003-2007. Int J Cardiol. 2010 Nov 19;145(2):242-244. doi: 10.1016/j.ijcard.2009.08.026. Epub 2009 Sep 15. PMID 19755203